CLINICAL TRIAL: NCT05011058
Title: An Open-Label, Phase 2 Trial of Nanatinostat in Combination With Valganciclovir in Patients With Epstein-Barr Virus-Positive (EBV+) Relapsed/Refractory Lymphomas
Brief Title: An Open-Label Phase 2 Trial of Nanatinostat Plus Valganciclovir in Patients With EBV+ Relapsed/Refractory Lymphomas
Acronym: NAVAL-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Viracta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VT3996-202
Record Dates: First submitted 2021-08-02; First posted 2021-08-18 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Epstein-Barr Virus Associated Lymphoma; EBV-Positive DLBCL, NOS; EBV-Related Non-Hodgkin Lymphoma; EBV Related PTCL, NOS; EBV-Related Hodgkin Lymphoma; EBV-Related PTLD; EBV-Related Lymphoproliferative Disorder
Keywords: Epstein-Barr virus (EBV); EBV-positive lymphomas; EBV-positive T-cell lymphoma; EBV-positive Hodgkin lymphoma; EBV-positive diffuse large B-cell lymphoma (DLBCL); EBV-positive extranodal natural killer/T-cell lymphoma; EBV-positive peripheral T-cell lymphoma (PTCL); EBV-positive post-transplant lymphoproliferative disorders
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic; Epstein-Barr Virus Infections | interventions — Valganciclovir

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm study utilizing a basket trial design.
  The study was terminated prematurely and did not reach its target enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nanatinostat with Valganciclovir (Experimental): Patients will receive nanatinostat 20 mg orally once daily, days 1-4 per week with valganciclovir 900 mg orally once daily.
  Up to 10 PTCL patients will receive nanatinostat 20 mg orally once daily, days 1-4 per week.
  Interventions: Drug: Nanatinostat in combination with valganciclovir

INTERVENTIONS:
Drug: Nanatinostat in combination with valganciclovir — Drug: Nanatinostat, 20 mg orally once daily, 4 days per week in 28 day cycles
  Drug: Valganciclovir, 900 mg orally once daily in 28 day cycles
  Other Names: VRx-3996 in combination with Valcyte

SUMMARY:
A Phase 2 study to evaluate the efficacy of nanatinostat in combination with valganciclovir in patients with relapsed/refractory EBV-positive lymphomas

DETAILED DESCRIPTION:
Patients with EBV-associated lymphomas have inferior outcomes with standard-of-care therapies compared to those with EBV-negative disease. Nanatinostat is a selective class I HDAC inhibitor which induces EBV lytic phase protein generation, activating (val)ganciclovir to its cytotoxic form. This open-label, multicenter, multinational, single-arm, Phase 2 basket study employs a Simon's 2-stage design to allow termination of enrollment into cohorts where treatment appears futile, and will include the following cohorts of patients with EBV+ relapsed/refractory lymphomas:

1. Diffuse large B-cell lymphoma (DLBCL)
2. Extranodal natural killer/T-cell lymphoma (ENKTL)
3. Peripheral T-cell lymphoma (PTCL), including angioimmunoblastic T-cell lymphoma (AITL) and PTCL not otherwise specified (PTCL-NOS)
4. Hodgkin lymphoma (HL)
5. Post-transplant lymphoproliferative disorders (PTLD)
6. Human immunodeficiency virus (HIV)-associated lymphomas (HIV-L)
7. EBV+ lymphomas other than the above

The study was terminated prematurely and did not reach its target enrollment.

ELIGIBILITY:
Key Inclusion Criteria:

* EBV+ DLBCL, NOS and PTCL, NOS, and AITL: Relapsed/refractory disease following 1 or more prior systemic therapy(ies) with curative intent.
* For EBV+ PTLD patients: Relapsed/refractory disease following 1 prior therapy and must have received at least 1 course of an anti-CD20 immunotherapy. For patients with EBV+ PTLD only, age 12 years and older and weighing greater than 40 kg (Adolescent, Adult, Older Adult) are allowed
* For other EBV+ relapsed/refractory lymphoma: Following at least 1 course of an anit-CD20 immunotherapy and at least 1 course of anthracycline-based chemotherapy (unless contraindicated)
* No available therapies in the opinion of the Investigator
* Not eligible for high-dose chemotherapy with allogeneic/autologous stem cell transplantation or CAR-T therapy
* Measurable disease per Cheson 2007
* ECOG performance status 0, 1, 2
* Adequate bone marrow function

Key Exclusion Criteria:

* Presence or history of CNS involvement by lymphoma
* Systemic anticancer therapy or CAR-T within 21 days
* Antibody (anticancer) agents within 28 days
* Less than 60 days from prior autologous hematopoietic stem cell or solid organ transplant
* Less than 90 days from prior allogeneic transplant.
* Daily corticosteroids (≥20 mg of prednisone or equivalent) within week prior to Cycle 1 Day 1
* Inability to take oral medication, malabsorption syndrome or any other gastrointestinal condition (nausea, diarrhea, vomiting) that may impact the absorption of nanatinostat and valganciclovir.
* Active infection requiring systemic therapy (excluding viral upper respiratory tract infections).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrel P Cohen, MD, PhD, Study Director — Viracta Therapeutics
Locations (62):
- United States (17):
  - The University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - City of Hope, Duarte, California
  - David Geffen School of Medicine - UCLA, Los Angeles, California
  - University of California Irvine, Orange, California
  - Scripps MD Anderson Cancer Center, San Diego, California
  - UCSF Hematology and Blood and Marrow Transplant, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Maryland Medical Center, Baltimore, Maryland
  - John Theurer Cancer Center: Hackensack Univeristy, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ohio State University: Wexner Medical Center, Columbus, Ohio
  - Sidney Kimmel Cancer Center - Jefferson Health, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (2):
  - Box Hill Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Brazil (5):
  - CEPEVILLE - Instituto Joinvilense de Hematologia e Oncologia, Joinville
  - Ruschel Medicina e Pesquisa Clinica, Rio de Janeiro
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
  - CIPE Centro Internacional de Pesquisa - AC Camargo Cancer Center, São Paulo
  - HCFMUSP - Hospital das Clínicas da Faculdade de Medicina Universidade de São Paulo, São Paulo
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
- France (6):
  - Institut Bergonié, Bordeaux, Aquitaine
  - Centre Hospitalier Universitaire Limoges, Limoges, Limousin
  - Hôpital Haut-Lévêque, Pessac, Nouvelle-Aquitaine
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite, Rhone-Alps
  - Henri Mondor University Hospital, Paris
  - Hôpital Universitaire Pitié Salpêtrière, Paris, Île-de-France Region
- Germany (2):
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Leipzig, Leipzig
- Hadassah Medical Center, Ein Kerem Hospital, Jerusalem, Israel
- Italy (9):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Centro di Riferimento Oncologico, Aviano, Pordenone
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant Orsola-Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Sarawak General Hospital / Hospital Umum Sarawak, Kuching, Malaysia
- Singapore (3):
  - National Cancer Centre Singapore, Singapore
  - Oncocare Cancer Center, Singapore
  - Singapore General Hospital, Singapore
- South Korea (2):
  - Gachon University Gil Medical Center, Incheon
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospitalet de Llobregat, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Jimenez Diaz Foundation University Hospital, Madrid
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan
- United Kingdom (3):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Derived] Haverkos B, Alpdogan O, Baiocchi R, Brammer JE, Feldman TA, Capra M, Brem EA, Nair S, Scheinberg P, Pereira J, Shune L, Joffe E, Young P, Spruill S, Katkov A, McRae R, Royston I, Faller DV, Rojkjaer L, Porcu P. Targeted therapy with nanatinostat and valganciclovir in recurrent EBV-positive lymphoid malignancies: a phase 1b/2 study. Blood Adv. 2023 Oct 24;7(20):6339-6350. doi: 10.1182/bloodadvances.2023010330. PMID 37530631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Epstein-Barr virus (EBV)-associated lymphoid malignancy were nonrandomly assigned to one of 7 cohorts defined in the Study Description module, except the first 20 patients with peripheral T-cell lymphoma were randomized (1:1) to receive either combination nanatinostat plus valganciclovir therapy or nanatinostat monotherapy.
  Up to 10 (Stage 1), up to 11 (Stage 2), and up to 120 (Expansion) patients were to be enrolled in each cohort depending on the number of responses observed.
Pre-assignment Details: Patients enrolled in the Peripheral T-Cell Lymphoma (Monotherapy) cohort who had stable disease at 6 weeks or disease progression at any time (confirmed by CT or MRI) were provided the option to cross over to receive combination therapy for the remainder of the study.
Groups:
- Diffuse Large B-Cell Lymphoma: Patients with relapsed or refractory EBV-positive diffuse large B-cell lymphoma treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD
- Extranodal Natural Killer/T-Cell Lymphoma: Patients with relapsed or refractory EBV-positive extranodal natural killer/T-cell lymphoma treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD
- Peripheral T-Cell Lymphoma (Combination Therapy): Patients with relapsed or refractory EBV-positive angioimmunoblastic T-cell lymphoma or peripheral T-cell lymphoma not otherwise specified treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD
- Peripheral T-Cell Lymphoma (Monotherapy): Patients with relapsed or refractory EBV-positive angioimmunoblastic T-cell lymphoma or peripheral T-cell lymphoma not otherwise specified treated with nanatinostat 20 mg QD on Days 1 to 4 per week
- Hodgkin Lymphoma: Patients with relapsed or refractory EBV-positive Hodgkin lymphoma treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD
- Post-Transplant Lymphoproliferative Disorders: Patients with relapsed or refractory EBV-positive post-transplant lymphoproliferative disorders treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD
- Human Immunodeficiency Virus-Associated Lymphomas: Patients with relapsed or refractory EBV-positive human immunodeficiency virus-associated lymphomas treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD
- Other EBV-Positive Lymphomas: Patients with relapsed or refractory EBV-positive lymphomas other than those from the other cohorts treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD
Period: Overall Study
Arm/Group | Diffuse Large B-Cell Lymphoma | Extranodal Natural Killer/T-Cell Lymphoma | Peripheral T-Cell Lymphoma (Combination Therapy) | Peripheral T-Cell Lymphoma (Monotherapy) | Hodgkin Lymphoma | Post-Transplant Lymphoproliferative Disorders | Human Immunodeficiency Virus-Associated Lymphomas | Other EBV-Positive Lymphomas
Started | 9 | 11 | 38 | 10 | 8 | 3 | 3 | 20
Stage 1 | 9 | 11 (More than 10 patients were enrolled in Stage 1 of the Extranodal Natural Killer/T-Cell Lymphoma cohort because the tenth and eleventh patients had signed informed consent concurrently.) | 10 | 10 | 8 | 3 | 3 | 20 (No more than 10 patients of a given lymphoma subtype were enrolled in Stage 1 of the Other EBV-Positive Lymphomas cohort.)
Stage 2 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0
Expansion | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0
Crossover (Crossover only applies to patients enrolled in the Peripheral T-Cell Lymphoma (Monotherapy) cohort who were subsequently provided the option to cross over to receive combination therapy.) | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Completed | 7 | 11 | 24 | 10 | 8 | 2 | 3 | 15
Not Completed | 2 | 0 | 14 | 0 | 0 | 1 | 0 | 5
Not completed — Sponsor Decision | 2 | 0 | 14 | 0 | 0 | 1 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diffuse Large B-Cell Lymphoma | Extranodal Natural Killer/T-Cell Lymphoma | Peripheral T-Cell Lymphoma (Combination Therapy) | Peripheral T-Cell Lymphoma (Monotherapy) | Hodgkin Lymphoma | Post-Transplant Lymphoproliferative Disorders | Human Immunodeficiency Virus-Associated Lymphomas | Other EBV-Positive Lymphomas | Total
Number analyzed (Participants) | 9 | 11 | 38 | 10 | 8 | 3 | 3 | 20 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14 | 4 | 7 | 2 | 3 | 9 | 53
  >=65 years | 3 | 3 | 24 | 6 | 1 | 1 | 0 | 11 | 49
Age, Continuous [Median (Full Range); unit: years] | 60 [21 to 82] | 53 [32 to 71] | 69 [47 to 85] | 69 [53 to 78] | 53.5 [23 to 69] | 50 [48 to 67] | 47 [46 to 57] | 64 [39 to 86] | 64 [21 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 19 | 2 | 4 | 0 | 0 | 6 | 37
  Male | 4 | 10 | 19 | 8 | 4 | 3 | 3 | 14 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 6 | 1 | 2 | 1 | 1 | 2 | 15
  Not Hispanic or Latino | 8 | 10 | 29 | 8 | 6 | 2 | 2 | 18 | 83
  Unknown or Not Reported | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 2 | 4 | 5 | 5 | 1 | 0 | 0 | 7 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3
  White | 7 | 3 | 29 | 4 | 6 | 1 | 3 | 11 | 64
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2 | 1 | 1 | 2 | 0 | 2 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 4
  United States | 0 | 4 | 12 | 1 | 4 | 2 | 1 | 6 | 30
  United Kingdom | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 3 | 7
  Spain | 1 | 0 | 9 | 1 | 2 | 0 | 0 | 0 | 13
  Canada | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 6
  South Korea | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Taiwan | 1 | 3 | 2 | 2 | 1 | 0 | 0 | 3 | 12
  Brazil | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 5
  Italy | 3 | 0 | 5 | 1 | 0 | 0 | 1 | 4 | 14
  Israel | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Australia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  France | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 6
  Germany | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Number (percentage) of patients with a best overall complete response (CR) or partial response (PR) according to the 2007 International Working Group (IWG) criteria, where CR included complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy with all lymph nodes and nodal masses having regressed on computed tomography to normal size, and PR included at least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses, no increase should have been observed in the size of other nodes, liver, or spleen, and splenic and hepatic nodules must have regressed by ≥ 50% in their SPD or, for single nodules, in the greatest transverse diameter.
Time Frame: Up to approximately 2 years
Population: Intent-to-Treat Analysis Set, defined as all patients who were enrolled into the trial regardless of whether or not they received study treatment.
  The study was not designed to make formal statistical comparisons of ORRs between cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-Cell Lymphoma | Extranodal Natural Killer/T-Cell Lymphoma | Peripheral T-Cell Lymphoma (Combination Therapy) | Peripheral T-Cell Lymphoma (Monotherapy) | Hodgkin Lymphoma | Post-Transplant Lymphoproliferative Disorders | Human Immunodeficiency Virus-Associated Lymphomas | Other EBV-Positive Lymphomas
Number analyzed (Participants) | 9 | 11 | 38 | 10 | 8 | 3 | 3 | 20
Participants | 0 | 0 | 11 | 1 | 0 | 0 | 0 | 2

2. Secondary Outcome: Duration of Response (DOR)
Description: Interval of time from date of first observed complete or partial response per 2007 International Working Group (IWG) criteria to the date of documented disease progression or death due to any cause, where disease progression is defined by 2007 IWG criteria as any new lesion or increase by ≥ 50% of previously involved sites from nadir. DOR was censored at the time of study withdrawal for hematopoietic stem cell transplant, or at the time of study termination, whichever was earlier, for patients whose disease was still in response.
Time Frame: Up to approximately 2 years
Population: Patients who achieved a CR or PR. The study was not designed to make formal statistical comparisons of DOR between cohorts.
Measure: Median (Full Range); unit: days
Arm/Group | Diffuse Large B-Cell Lymphoma | Extranodal Natural Killer/T-Cell Lymphoma | Peripheral T-Cell Lymphoma (Combination Therapy) | Peripheral T-Cell Lymphoma (Monotherapy) | Hodgkin Lymphoma | Post-Transplant Lymphoproliferative Disorders | Human Immunodeficiency Virus-Associated Lymphomas | Other EBV-Positive Lymphomas
Number analyzed (Participants) | 0 | 0 | 11 | 1 | 0 | 0 | 0 | 2
days |  |  | 98 [29 to 340] | 43 [43 to 43] |  |  |  | 163.5 [86 to 241]

3. Secondary Outcome: Time to Next Anti-Lymphoma Treatment (TTNLT)
Description: Interval of time from the start of study drug treatment to the date of next anti-lymphoma treatment (including chemotherapy, radiotherapy, radioimmunotherapy, or immunotherapy).
Time Frame: Up to approximately 3 years
Population: The clinical trial was terminated before the outcome measure data were collected (data export from the clinical database just prior to study termination retrieved from data manager files contained data listings to support determinations of other secondary efficacy outcome measures but not post-treatment anticancer therapy regimen dates to support TTNLT determination, and investigation into the cause of these uncollected data was preempted by sponsor company closure soon after study termination).
Arm/Group | Diffuse Large B-Cell Lymphoma | Extranodal Natural Killer/T-Cell Lymphoma | Peripheral T-Cell Lymphoma (Combination Therapy) | Peripheral T-Cell Lymphoma (Monotherapy) | Hodgkin Lymphoma | Post-Transplant Lymphoproliferative Disorders | Human Immunodeficiency Virus-Associated Lymphomas | Other EBV-Positive Lymphomas
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Time to Progression (TTP)
Description: Interval of time from the start of study drug treatment to the date of disease progression, where disease progression is defined by 2007 IWG criteria as any new lesion or increase by ≥ 50% of previously involved sites from nadir. TTP was censored at the time of study withdrawal for hematopoietic stem cell transplant, at the time of study treatment withdrawal (or at the time of crossover from monotherapy to combination therapy), or at the time of study termination, whichever was earliest, for patients without reported disease progression.
Time Frame: Up to approximately 3 years
Population: Intent-to-Treat Analysis Set, defined as all patients who were enrolled into the trial regardless of whether or not they received study treatment.
  The study was not designed to make formal statistical comparisons of TTP between cohorts.
Measure: Median (Full Range); unit: days
Arm/Group | Diffuse Large B-Cell Lymphoma | Extranodal Natural Killer/T-Cell Lymphoma | Peripheral T-Cell Lymphoma (Combination Therapy) | Peripheral T-Cell Lymphoma (Monotherapy) | Hodgkin Lymphoma | Post-Transplant Lymphoproliferative Disorders | Human Immunodeficiency Virus-Associated Lymphomas | Other EBV-Positive Lymphomas
Number analyzed (Participants) | 9 | 11 | 38 | 10 | 8 | 3 | 3 | 20
days | 81 [29 to 165] | 100 [23 to 260] | 124 [14 to 410] | 95 [32 to 136] | 77.5 [64 to 127] | 79 [36 to 351] | 108 [64 to 282] | 95.5 [35 to 311]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: Interval of time from the start of study drug treatment to the date of first documented disease progression (defined by 2007 IWG criteria as any new lesion or increase by ≥ 50% of previously involved sites from nadir), initiation of new antineoplastic therapy, or death from any cause, whichever occurred first. PFS was censored at the time of study withdrawal for hematopoietic stem cell transplant, at the time of study treatment withdrawal (or at the time of crossover from monotherapy to combination therapy), or at the time of study termination, whichever was earliest, for patients without reported disease progression or death.
Time Frame: Up to approximately 3 years
Population: Intent-to-Treat Analysis Set, defined as all patients who were enrolled into the trial regardless of whether or not they received study treatment.
  The study was not designed to make formal statistical comparisons of PFS between cohorts.
Measure: Median (Full Range); unit: days
Arm/Group | Diffuse Large B-Cell Lymphoma | Extranodal Natural Killer/T-Cell Lymphoma | Peripheral T-Cell Lymphoma (Combination Therapy) | Peripheral T-Cell Lymphoma (Monotherapy) | Hodgkin Lymphoma | Post-Transplant Lymphoproliferative Disorders | Human Immunodeficiency Virus-Associated Lymphomas | Other EBV-Positive Lymphomas
Number analyzed (Participants) | 9 | 11 | 38 | 10 | 8 | 3 | 3 | 20
days | 81 [29 to 165] | 110 [23 to 517] | 124 [14 to 410] | 95 [32 to 171] | 82 [64 to 313] | 79 [36 to 351] | 108 [64 to 282] | 95.5 [35 to 311]

6. Secondary Outcome: Overall Survival (OS)
Description: Interval of time from the start of study drug treatment to the date of death for any reason. OS was censored at the time of study withdrawal or study termination, whichever was earlier, for patients without reported death.
Time Frame: Up to approximately 3 years
Population: Intent-to-Treat Analysis Set, defined as all patients who were enrolled into the trial regardless of whether or not they received study treatment.
  The study was not designed to make formal statistical comparisons of OS between cohorts.
Measure: Median (Full Range); unit: days
Arm/Group | Diffuse Large B-Cell Lymphoma | Extranodal Natural Killer/T-Cell Lymphoma | Peripheral T-Cell Lymphoma (Combination Therapy) | Peripheral T-Cell Lymphoma (Monotherapy) | Hodgkin Lymphoma | Post-Transplant Lymphoproliferative Disorders | Human Immunodeficiency Virus-Associated Lymphomas | Other EBV-Positive Lymphomas
Number analyzed (Participants) | 9 | 11 | 38 | 10 | 8 | 3 | 3 | 20
days | 131 [29 to 242] | 243 [35 to 517] | 221 [14 to 730] | 155 [41 to 611] | 570.5 [64 to 1000] | 171 [36 to 351] | 108 [76 to 296] | 167.5 [35 to 513]

7. Secondary Outcome: Number (Percentage) of Participants With Adverse Events (AEs)
Description: Number (percentage) of patients experiencing at least one treatment-emergent adverse event, defined as those untoward medical events with onset after the first dose of study drug or existing events that worsened after the first dose during the study
Time Frame: Up to approximately 2 years
Population: Safety Analysis Set, defined as all enrolled patients who received at least 1 dose of study treatment.
  The study was not designed to make formal statistical comparisons of AE numbers (percentages) between cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-Cell Lymphoma | Extranodal Natural Killer/T-Cell Lymphoma | Peripheral T-Cell Lymphoma (Combination Therapy) | Peripheral T-Cell Lymphoma (Monotherapy) | Hodgkin Lymphoma | Post-Transplant Lymphoproliferative Disorders | Human Immunodeficiency Virus-Associated Lymphomas | Other EBV-Positive Lymphomas
Number analyzed (Participants) | 9 | 11 | 38 | 10 | 8 | 3 | 3 | 20
Participants | 9 | 10 | 32 | 10 | 7 | 3 | 3 | 17

8. Secondary Outcome: Pharmacokinetic (PK) Parameter - Time to Maximum Plasma Concentration [Tmax]
Description: Defined as the time required to reach peak plasma concentration [Cmax] after study drug administration
Time Frame: Cycle 1 Day 1 and Cycle 6 Day 1 at pre-dose and 1, 2, 4, and 6 hours post-dose (each cycle was 28 days)
Population: Defined as all patients (pts) who received at least 1 dose of study drug on Cycle 1 Day 1 and had at least 1 valid PK concentration. Tmax data were previously generated for subset of 50 pts, 4 of whom reached Cycle 6 at time of analysis. As prespecified by the analysis plan, combination therapy cohorts were combined since Tmax for small molecules should not be affected by lymphoma subtype. PK samples from remaining pts were not tested due to sponsor company closure soon after study termination.
Measure: Median (Full Range); unit: hours
Groups:
- Combination Therapy (EBV-Associated Lymphoid Malignancy): Patients with relapsed or refractory EBV-positive lymphoma or lymphoproliferative disorder treated with nanatinostat 20 mg once daily (QD) on Days 1 to 4 per week and valganciclovir 900 mg QD
- Monotherapy (EBV-Positive Peripheral T-Cell Lymphoma): Patients with relapsed or refractory EBV-positive angioimmunoblastic T-cell lymphoma or peripheral T-cell lymphoma not otherwise specified treated with nanatinostat 20 mg QD on Days 1 to 4 per week
Arm/Group | Combination Therapy (EBV-Associated Lymphoid Malignancy) | Monotherapy (EBV-Positive Peripheral T-Cell Lymphoma)
Number analyzed (Participants) | 40 | 10
hours
  Nanatinostat (Cycle 1 Day 1) | 2 [1 to 6] | 2 [1 to 4]
  Nanatinostat (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  Nanatinostat (Cycle 6 Day 1) | 2 [1 to 6] |
  M1 Metabolite (Cycle 1 Day 1) | 6 [2 to 6] | 5 [2 to 6]
  M1 Metabolite (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  M1 Metabolite (Cycle 6 Day 1) | 5 [2 to 6] |
  M2 Metabolite (Cycle 1 Day 1) | 4 [1 to 6] | 2 [1 to 6]
  M2 Metabolite (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  M2 Metabolite (Cycle 6 Day 1) | 4 [1 to 6] |
  Ganciclovir (Cycle 1 Day 1): number analyzed (Participants) | 40 | 0
  Ganciclovir (Cycle 1 Day 1) | 2 [1 to 6] |
  Ganciclovir (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  Ganciclovir (Cycle 6 Day 1) | 2 [2 to 2] |

9. Secondary Outcome: Pharmacokinetic (PK) Parameter - Maximum Plasma Concentration [Cmax]
Description: Defined as the peak plasma concentration [Cmax] after study drug administration
Time Frame: Cycle 1 Day 1 and Cycle 6 Day 1 at pre-dose and 1, 2, 4, and 6 hours post-dose (each cycle was 28 days)
Population: Defined as all patients (pts) who received at least 1 dose of study drug on Cycle 1 Day 1 and had at least 1 valid PK concentration. Cmax data were previously generated for subset of 50 pts, 4 of whom reached Cycle 6 at time of analysis. As prespecified by the analysis plan, combination therapy cohorts were combined since Cmax for small molecules should not be affected by lymphoma subtype. PK samples from remaining pts were not tested due to sponsor company closure soon after study termination.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Combination Therapy (EBV-Associated Lymphoid Malignancy) | Monotherapy (EBV-Positive Peripheral T-Cell Lymphoma)
Number analyzed (Participants) | 40 | 10
ng/mL
  Nanatinostat (Cycle 1 Day 1) | 116 (68.9) | 105 (83.0)
  Nanatinostat (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  Nanatinostat (Cycle 6 Day 1) | 134 (121.3) |
  M1 Metabolite (Cycle 1 Day 1) | 435 (49.6) | 393 (48.3)
  M1 Metabolite (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  M1 Metabolite (Cycle 6 Day 1) | 427 (64.6) |
  M2 Metabolite (Cycle 1 Day 1) | 75.1 (56.5) | 65.8 (64.3)
  M2 Metabolite (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  M2 Metabolite (Cycle 6 Day 1) | 82.8 (79.0) |
  Ganciclovir (Cycle 1 Day 1): number analyzed (Participants) | 40 | 0
  Ganciclovir (Cycle 1 Day 1) | 6350 (35.7) |
  Ganciclovir (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  Ganciclovir (Cycle 6 Day 1) | 5390 (59.6) |

10. Secondary Outcome: Pharmacokinetic Parameter - Area Under the Plasma Concentration-Time Curve [AUC0-t]
Description: Defined as the area under the concentration-time curve from time 0 to the last measurable plasma concentration
Time Frame: Cycle 1 Day 1 and Cycle 6 Day 1 at pre-dose and 1, 2, 4, and 6 hours post-dose (each cycle was 28 days)
Population: Defined as all patients (pts) who received at least 1 dose of study drug on Cycle 1 Day 1 and had at least 1 valid PK concentration. AUC0-t data were previously generated for subset of 50 pts, 4 of whom reached Cycle 6 at time of analysis. As prespecified by the analysis plan, combination therapy cohorts were combined since AUC for small molecules should not be affected by lymphoma subtype. PK samples from remaining pts were not tested due to sponsor company closure soon after study termination.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Combination Therapy (EBV-Associated Lymphoid Malignancy) | Monotherapy (EBV-Positive Peripheral T-Cell Lymphoma)
Number analyzed (Participants) | 40 | 10
ng*h/mL
  Nanatinostat (Cycle 1 Day 1) | 284 (46.9) | 241 (59.3)
  Nanatinostat (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  Nanatinostat (Cycle 6 Day 1) | 291 (101.2) |
  M1 Metabolite (Cycle 1 Day 1) | 1470 (70.6) | 1410 (56.8)
  M1 Metabolite (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  M1 Metabolite (Cycle 6 Day 1) | 3750 (42.2) |
  M2 Metabolite (Cycle 1 Day 1) | 263 (71.9) | 248 (66.2)
  M2 Metabolite (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  M2 Metabolite (Cycle 6 Day 1) | 335 (168.2) |
  Ganciclovir (Cycle 1 Day 1): number analyzed (Participants) | 40 | 0
  Ganciclovir (Cycle 1 Day 1) | 21600 (34.9) |
  Ganciclovir (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  Ganciclovir (Cycle 6 Day 1) | 33400 (20.4) |

11. Secondary Outcome: Pharmacokinetic (PK) Parameter - Half-Life [t1/2]
Description: Defined as the time required to reduce plasma concentration by 50% after study drug administration
Time Frame: Cycle 1 Day 1 and Cycle 6 Day 1 at pre-dose and 1, 2, 4, and 6 hours post-dose (each cycle was 28 days)
Population: Defined as all patients who received at least 1 dose of study drug on Cycle 1 Day 1 and had at least 2 valid PK concentrations in the terminal elimination phase. This stricter requirement explains why, for example, the overall number analyzed for t1/2 (ie, 16) is less than the overall number analyzed for the other PK parameters (ie, 50). As prespecified by the analysis plan, combination therapy cohorts were combined since t1/2 for small molecules should not be affected by lymphoma subtype.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Combination Therapy (EBV-Associated Lymphoid Malignancy) | Monotherapy (EBV-Positive Peripheral T-Cell Lymphoma)
Number analyzed (Participants) | 12 | 4
hours
  Nanatinostat (Cycle 1 Day 1) | 1.52 (0.464) | 2.17 (0.503)
  Nanatinostat (Cycle 6 Day 1): number analyzed (Participants) | 1 | 0
  Nanatinostat (Cycle 6 Day 1) | 1.21 (0) |
  Ganciclovir (Cycle 1 Day 1): number analyzed (Participants) | 9 | 0
  Ganciclovir (Cycle 1 Day 1) | 3.41 (1.34) |
  Ganciclovir (Cycle 6 Day 1): number analyzed (Participants) | 4 | 0
  Ganciclovir (Cycle 6 Day 1) | 5.31 (2.36) |

12. Other Pre Specified Outcome: Objective Response Rate (ORR) by Study Milestone in the Peripheral T-Cell Lymphoma (Combination Therapy) Cohort That Enrolled Patients Beyond Stage 1 or in the Peripheral T-Cell Lymphoma (Monotherapy) Cohort Who Crossed Over to Receive Combination Therapy
Description: as for outcome 1
Time Frame: Up to approximately 2 years
Population: Intent-to-Treat Analysis Set, defined as all patients who were enrolled into the trial regardless of whether or not they received study treatment.
  The sum of the Overall Number of Participants Analyzed across all subgroups (ie, 57) additionally includes pre-specified ORR analyses in a subset of 14 patients in the Peripheral T-Cell Lymphoma (Combination Therapy) cohort previously treated with only 1 line of anti-lymphoma therapy.
Measure: Count of Participants; unit: Participants
Groups:
- Stage 1 (Peripheral T-Cell Lymphoma): Patients with relapsed or refractory EBV-positive angioimmunoblastic T-cell lymphoma or peripheral T-cell lymphoma not otherwise specified treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD in the first stage of the study
- Stage 1 (Peripheral T-Cell Lymphoma - Second Line): Patients with second-line relapsed or refractory EBV-positive angioimmunoblastic T-cell lymphoma or peripheral T-cell lymphoma not otherwise specified treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD in the first stage of the study
- Stage 2 (Peripheral T-Cell Lymphoma): Patients with relapsed or refractory EBV-positive angioimmunoblastic T-cell lymphoma or peripheral T-cell lymphoma not otherwise specified treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD in the second stage of the study
- Stage 2 (Peripheral T-Cell Lymphoma - Second Line): Patients with second-line relapsed or refractory EBV-positive angioimmunoblastic T-cell lymphoma or peripheral T-cell lymphoma not otherwise specified treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD in the second stage of the study
- Expansion (Peripheral T-Cell Lymphoma): Patients with relapsed or refractory EBV-positive angioimmunoblastic T-cell lymphoma or peripheral T-cell lymphoma not otherwise specified treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD in the expansion stage of the study
- Expansion (Peripheral T-Cell Lymphoma - Second Line): Patients with second-line relapsed or refractory EBV-positive angioimmunoblastic T-cell lymphoma or peripheral T-cell lymphoma not otherwise specified treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD in the expansion stage of the study
- Crossover (Peripheral T-Cell Lymphoma): Patients with relapsed or refractory EBV-positive angioimmunoblastic T-cell lymphoma or peripheral T-cell lymphoma not otherwise specified treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD after having been treated with nanatinostat 20 mg QD on Days 1 to 4 per week without response in the monotherapy cohort
Arm/Group | Stage 1 (Peripheral T-Cell Lymphoma) | Stage 1 (Peripheral T-Cell Lymphoma - Second Line) | Stage 2 (Peripheral T-Cell Lymphoma) | Stage 2 (Peripheral T-Cell Lymphoma - Second Line) | Expansion (Peripheral T-Cell Lymphoma) | Expansion (Peripheral T-Cell Lymphoma - Second Line) | Crossover (Peripheral T-Cell Lymphoma)
Number analyzed (Participants) | 10 | 5 | 11 | 4 | 17 | 5 | 5
Participants | 5 | 5 | 2 | 1 | 4 | 1 | 2

13. Other Pre Specified Outcome: Duration of Response (DOR) by Study Milestone in the Peripheral T-Cell Lymphoma (Combination Therapy) Cohort That Enrolled Patients Beyond Stage 1 or in the Peripheral T-Cell Lymphoma (Monotherapy) Cohort Who Crossed Over to Receive Combination Therapy
Description: as for outcome 2
Time Frame: Up to approximately 2 years
Population: Patients who achieved a CR or PR
Measure: Median (Full Range); unit: days
Groups:
- Peripheral T-Cell Lymphoma (Crossover): Patients with relapsed or refractory EBV-positive angioimmunoblastic T-cell lymphoma or peripheral T-cell lymphoma not otherwise specified treated with nanatinostat 20 mg QD on Days 1 to 4 per week and valganciclovir 900 mg QD after having been treated with nanatinostat 20 mg QD on Days 1 to 4 per week without response in the monotherapy cohort
Arm/Group | Stage 1 (Peripheral T-Cell Lymphoma) | Stage 1 (Peripheral T-Cell Lymphoma - Second Line) | Stage 2 (Peripheral T-Cell Lymphoma) | Stage 2 (Peripheral T-Cell Lymphoma - Second Line) | Expansion (Peripheral T-Cell Lymphoma) | Expansion (Peripheral T-Cell Lymphoma - Second Line) | Peripheral T-Cell Lymphoma (Crossover)
Number analyzed (Participants) | 5 | 5 | 2 | 1 | 4 | 1 | 2
days | 86 [36 to 340] | 86 [36 to 340] | 125 [29 to 221] | 29 [29 to 29] | 99 [73 to 126] | 73 [73 to 73] | 192 [79 to 305]

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years for All-Cause Mortality; Up to approximately 2 years for Serious Adverse Events and Other (Not Including Serious) Adverse Events
Arm/Group | Diffuse Large B-Cell Lymphoma | Extranodal Natural Killer/T-Cell Lymphoma | Peripheral T-Cell Lymphoma (Combination Therapy) | Peripheral T-Cell Lymphoma (Monotherapy) | Peripheral T-Cell Lymphoma (Crossover) | Hodgkin Lymphoma | Post-Transplant Lymphoproliferative Disorders | Human Immunodeficiency Virus-Associated Lymphomas | Other EBV-Positive Lymphomas
All-Cause Mortality (participants affected / at risk) | 3/9 | 9/11 | 9/38 | 4/10 | 2/5 | 3/8 | 1/3 | 1/3 | 8/20
Serious Adverse Events (participants affected / at risk) | 3/9 | 7/11 | 9/38 | 5/10 | 3/5 | 2/8 | 3/3 | 2/3 | 10/20
Other Adverse Events (participants affected / at risk) | 9/9 | 10/11 | 32/38 | 10/10 | 5/5 | 7/8 | 3/3 | 3/3 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-Cell Lymphoma (N=9) | Extranodal Natural Killer/T-Cell Lymphoma (N=11) | Peripheral T-Cell Lymphoma (Combination Therapy) (N=38) | Peripheral T-Cell Lymphoma (Monotherapy) (N=10) | Peripheral T-Cell Lymphoma (Crossover) (N=5) | Hodgkin Lymphoma (N=8) | Post-Transplant Lymphoproliferative Disorders (N=3) | Human Immunodeficiency Virus-Associated Lymphomas (N=3) | Other EBV-Positive Lymphomas (N=20)
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 4
Sepsis (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 3 | 1 | 2 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-Cell Lymphoma (N=9) | Extranodal Natural Killer/T-Cell Lymphoma (N=11) | Peripheral T-Cell Lymphoma (Combination Therapy) (N=38) | Peripheral T-Cell Lymphoma (Monotherapy) (N=10) | Peripheral T-Cell Lymphoma (Crossover) (N=5) | Hodgkin Lymphoma (N=8) | Post-Transplant Lymphoproliferative Disorders (N=3) | Human Immunodeficiency Virus-Associated Lymphomas (N=3) | Other EBV-Positive Lymphomas (N=20)
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 7 | 5 | 3 | 4 | 0 | 2 | 7
Nausea (Gastrointestinal disorders) | 1 | 7 | 12 | 1 | 1 | 4 | 1 | 1 | 5
Neutrophil count decreased (Investigations) | 3 | 4 | 9 | 3 | 3 | 3 | 1 | 1 | 7
Fatigue (General disorders) | 2 | 4 | 8 | 4 | 1 | 2 | 2 | 2 | 7
Pyrexia (General disorders) | 2 | 6 | 12 | 3 | 1 | 1 | 1 | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4 | 9 | 5 | 0 | 3 | 0 | 0 | 5
Platelet count decreased (Investigations) | 2 | 4 | 8 | 4 | 2 | 1 | 0 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 6 | 3 | 1 | 3 | 1 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5 | 0 | 0 | 3 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 4 | 4 | 0 | 0 | 1 | 1 | 0 | 3
White blood cell decreased (Investigations) | 1 | 1 | 4 | 2 | 2 | 2 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 5 | 1 | 0 | 1 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1 | 5 | 0 | 1 | 2 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 2 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 3
Asthenia (General disorders) | 1 | 0 | 3 | 1 | 0 | 2 | 0 | 1 | 2
COVID-19 (Infections and infestations) | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0 | 2 | 1 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 2 | 3 | 0 | 1 | 1 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
The study was terminated prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT05011058/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT05011058/SAP_001.pdf